CLINICAL TRIAL: NCT02935608
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of BIIB074 in Subjects With Neuropathic Pain From Lumbosacral Radiculopathy
Brief Title: Study to Evaluate the Efficacy and Safety of BIIB074 in Neuropathic Pain From Lumbosacral Radiculopathy
Acronym: RELAY-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1014802-203; 2015-004775-78 (EudraCT Number)
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Lumbosacral Radiculopathy
MeSH Terms: interventions — vixotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BIIB074 high dose (Experimental): Administered twice daily (BID)
  Interventions: Drug: BIIB074
- BIIB074 low dose (Experimental): Administered BID
  Interventions: Drug: BIIB074
- Placebo (Placebo Comparator): Placebo administered BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB074 — Administered as specified in the treatment arm
  Other Names: CNV1014802
  Arms: BIIB074 high dose; BIIB074 low dose
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of two dose regimens of BIIB074 on neuropathic pain in participants with pain from lumbosacral radiculopathy (PLSR). Secondary objectives are to evaluate the efficacy of 2 dose regimens of BIIB074 on additional neuropathic pain measures and assessments of low back pain, disability, and quality of life; To investigate the safety and tolerability of 2 dose regimens of BIIB074 and To characterize the pharmacokinetics (PK) of BIIB074 in this population.

DETAILED DESCRIPTION:
This study was previously posted by Convergence Pharmaceuticals, Ltd., which has been acquired by Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Has body weight ≥50 kg for men and ≥45 kg for women
* Must have diagnosis of neuropathic PLSR
* Has duration of neuropathic (leg) pain of at least 6 months before Screening
* Has an intensity of ≥4 and ≤9 on the Numerical Rating Scale based on a paper-based question at Screening and on Day 1 that asks for the average pain intensity of neuropathic (leg) pain due to PLSR over the last week

Key Exclusion Criteria:

* Has planned surgical intervention for PLSR within the duration of the study. (Subjects with persistent radicular pain after prior surgery are eligible.)
* Has a history of peripheral neuropathy (e.g., due to diabetes, alcohol consumption, other causes, or idiopathic) or evidence of peripheral neuropathy upon neurological examination
* Has a history or risk of seizures or a history of epilepsy, clinically significant head injury, or related neurological disorders

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 14 in the weekly average of the daily neuropathic pain score on the 11-point Pain Intensity Numerical Rating Scale (PI-NRS) | Week 14
  Participants will be asked every evening to rate their overall neuropathic pain for the last 24-hour period. PI-NRS is an 11-point pain intensity numerical rating scale (PI-NRS), where 0=no pain and 10=pain as bad as you can imagine.

SECONDARY OUTCOMES:
50% neuropathic daily pain reduction response | At Week 14
  Response is defined as a ≥50% reduction in the weekly average of the daily neuropathic pain score from Baseline (Week 2) to Week 14.
30% neuropathic daily pain reduction response | At Week 14
  Response is defined as a ≥30% reduction in the weekly average of the daily neuropathic pain score from Baseline to Week 14.
Change from Baseline to Week 14 in the weekly average of the daily neuropathic pain score at each visit | Week 14
Change from Baseline to Week 14 in weekly average of the daily pain score for low back pain | Week 14
  Participants will be asked every evening to rate their overall low back pain for the last 24-hour period
Number of Patient Global Impression of Change (PGIC) responders | At Week 14
  PGIC is a 7-point, self-report scale depicting a participant's rating of overall improvement. Participants rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Change from Baseline to Week 14 on the Oswestry Disability Index | Week 14
  This is a 10-item questionnaire that evaluates how back (or leg) pain affects the ability to manage in everyday life. Each question is rated on a 5 point scale with higher scores indicating higher level of pain.
Change from Baseline to Week 14 in the weekly average of daily sleep score as assessed by the Sleep Numerical Rating Scale (S-NRS) | Week 14
  Participants will be asked every morning to rate on the 11-point S-NRS how leg pain interfered with their sleep quality, where 0=no pain and 10=Pain completely interfered with sleep.
Change from Baseline to Week 14 in the Brief Pain Inventory (BPI)- Interference index | Week 14
  BPI Interference Index is an 11-point numeric rating scale (0 - no interference to 10 - interferes completely) to assess pain-related interference in 7 areas: general activity, mood, walking ability, normal work, including outside the home and housework, relations with other people, enjoyment of life and sleep.
Change from Baseline to Week 14 in the BPI-Pain index | Week 14
  BPI- Pain Index for pain intensity is used to assess potential pain quality descriptors that may describe participants' pain on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
Change from Baseline to Week 14 on the EuroQoL 5-Dimension 5-Level Questionnaire (EQ-5D-5L) health index | Week 14
  The EQ-5D-3L is a standardized instrument for use as a measure of health outcome. It is a health questionnaire that consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.
Change from Baseline to Week 14 in Short Form 36 Questionnaire (SF-36) | Week 14
  SF-36 is a self-administered, generic health status questionnaire consisting of 36 questions that measure 8 health concepts: physical functioning, role limitations due to physical problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional problems and mental health.
Amount of rescue medication used per day | Day 1 to Week 15
Number of participants experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 15
Number of participants with clinically significant vital sign abnormalities | Up to Week 15
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities | Up to Week 15
Number of participants with clinically significant laboratory assessment abnormalities | Up to Week 15
Safety and Tolerability as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Week 15
  C-SSRS is a suicidal ideation rating used to evaluate suicidality in children ages 12 and up. It rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent."
Area under the concentration-time curve over the dosing period (AUCtau) at steady state | 30 min prior to dosing up to 8 hours post dose
Maximum concentration (Cmax) | 30 min prior to dosing up to 8 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (39):
- Research Site, Klagenfurt, Austria
- Research Site, Leuven, Belgium
- Bulgaria (4):
  - Research Site, Blagoevgrad
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Veliko Tarnovo
- Czechia (8):
  - Research Site, Beroun
  - Research Site, Choceň
  - Research Site, Litoměřice
  - Research Site, Litomyšl
  - Research Site, Ostrava
  - Research Site, Prachatice
  - Research Site, Prague
  - Research Site, Zlín
- Research Site, Paris, France
- Research Site, Tbilisi, Georgia
- Italy (2):
  - Research Site, Milan
  - Research Site, Rome
- Latvia (2):
  - Research Site, Liepāja
  - Research Site, Riga
- Research Site, Nieuwegein, Netherlands
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
- Research Site, Belgrade, Serbia
- Slovakia (6):
  - Research Site, Banská Bystrica
  - Research Site, Dolný Kubín
  - Reasearch Site, Dubnica nad Váhom
  - Research Site, Krompachy
  - Research Site, Pruské
  - Research Site, Spišská Nová Ves
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Elche
  - Research Site, Granada
  - Research Site, Madrid
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, Edinburgh
  - Research Site, Liverpool
  - Research Site, London